CLINICAL TRIAL: NCT03241966
Title: Perception, Cognition, and Gait in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Alice Cronin-Golomb, Director of Vision and Cognition Laboratory, Boston University Charles River Campus
Other Study IDs: 1204E
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Online Study; Quality of Life; Activities of Daily Living; Perception; Cognition; Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with Parkinson's Disease: Individuals diagnosed with idiopathic Parkinson's disease without dementia.
- Informant: Family member, spouse, significant other, caregiver, or other close associate of someone with Parkinson's disease.

SUMMARY:
The investigators are examining how aspects of daily function are perceived in persons with PD and in those who interact with them on a regular basis. If eligible, participants will receive a set of online questionnaires by email. The questionnaires will take about 1 hour to complete, and can be done at the participant's convenience. The investigators are looking for volunteers who have a diagnosis of Parkinson's disease without dementia (age 40 or older and proficient English speakers). If a spouse, family member, significant other or other close associate is available (age 18 or older, proficient English speakers), the investigators will send them questionnaires as well. There is no monetary or other compensation for this study. For more information, please contact the Vision and Cognition Laboratory at vcognition@gmail.com or 617-358-1377.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease without dementia OR close associate of someone with Parkinson's disease
* 40 years or older
* Proficient English speaker
* Access to a computer
* 8+ years of education

Exclusion Criteria:

* Co-existing active neoplasm, serious cardiac disease, other serious chronic medical illness
* Prior intracranial surgery
* History of traumatic brain injury
* Psychiatric or neurological diagnoses other than Parkinson's disease
* History of alcoholism or other drug abuse
* History of treatment with electroshock therapy

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are accepted regardless of location, community, clinic, etc.
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Questionnaire (PDQ-39) | Within 24 hours of starting the study
  Measures the health status of Parkinson's disease patients and the impact the disease has on their aspects of daily living. There are 39 items.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Cronin-Golomb, Ph.D., Principal Investigator — Boston University
Locations (1):
- Vision and Cognition Laboratory at Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No